CLINICAL TRIAL: NCT02952729
Title: A Phase 1b, First-in-Human, Dose Escalation and Expansion Study of XMT-1522 in Patients With Advanced Breast Cancer and Other Advanced Tumors Expressing HER2
Brief Title: Study of Antibody Drug Conjugate in Patients With Advanced Breast Cancer Expressing HER2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mersana Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMT-1522-1
Record Dates: First submitted 2016-10-27; First posted 2016-11-02 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Advanced Breast Cancer; Advanced Nonsmall Cell Lung Cancer; Advanced Gastric Cancer
MeSH Terms: interventions — XMT-1522

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation and Confirmation (Experimental): XMT-1522 treatment will administered in groups of patients who will receive doses that increase over time. Once the maximum tolerated dose or recommended Phase 2 dose is achieved, new groups of patients will receive XMT-1522 at this fixed dose.
  Interventions: Drug: XMT-1522

INTERVENTIONS:
Drug: XMT-1522 — one intravenous dose administered in-clinic every 21 days

SUMMARY:
This Phase 1b trial is an open label, multi-center study of XMT-1522 administered as an intravenous infusion once every three weeks. The dose escalation part of the study will establish the maximum tolerated dose or recommended Phase 2 dose for in patients with advanced breast cancer and either a HER2 immunohistochemistry (IHC) score of at least 1+ using a validated IHC assay or with evidence of HER2 amplification. Patients with HER2 positive (by IHC or amplification) gastric cancer or nonsmall cell lung cancer may also be eligible for participation in dose escalation. Upon completion of dose escalation, the cohort expansion segment of the study will consist of four parallel cohorts of different patients groups to confirm the maximum tolerated dose or the recommended Phase 2 dose and estimate the objective response in each of the patient populations.

DETAILED DESCRIPTION:
The dose escalation segment of the study utilizes a 3+3 design. Initially, 3 patients will be dosed at each dose level. The first 3-week cycle of treatment constitutes the dose limiting toxicity (DLT) evaluation period. If none of the 3 patients experience a DLT during the evaluation period and the Safety Review Committee agrees this was a reasonably well tolerated dose, 3 patients will be enrolled at the next dose level. However, in the event of 1 DLT, 3 additional patients will be enrolled at the same dose level. Any dose level with 2 or more DLTs will be considered to have exceeded the maximum tolerated dose and subsequent patients will be enrolled at lower dose levels. After the first cycle, patients may continue to receive XMT-1522 until disease progression as long as the drug is well-tolerated and patients continue to derive clinical benefit in the opinion of the Investigator.

After completion of the dose escalation, the expansion segment will enroll the patients with the following kinds of cancer:

* Cohort 1: Advanced breast cancer, HER2 IHC 1+, or HER2 IHC 2+ without HER2 gene amplification
* Cohort 2: Advanced breast cancer, HER2-positive, who have received prior ado-trastuzumab emtansine
* Cohort 3: Advanced gastric cancer, HER2-positive, who have received prior trastuzumab
* Cohort 4: Advanced non-small cell lung cancer, HER2 IHC 2+ or 3+, any HER2 gene amplification or mutation status

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease via RECIST
* Resolution of all toxic side effects from prior oncology treatments
* Adequate organ function as measured by various blood parameters
* Not pregnant or lactating, willing to prevent pregnancy while on study and for 6 months after the last dose of XMT-1522
* Histologically or cytologically confirmed adenocarcinoma of the breast with unresectable locally advanced disease, or metastatic disease and HER2 IHC 1+ or 2+ OR
* Histologically or cytologically confirmed adenocarcinoma of the breast with unresectable locally advanced disease, or metastatic disease and HER2 IHC 3+ or positive for HER2 gene amplification
* Progressed following all standard of care therapies for advanced breast cancer. OR
* Histologically or cytologically confirmed locally advanced or metastatic gastric cancer and HER2 IHC 3+ or positive for HER2 gene amplification OR
* Histologically or cytologically confirmed Stage IIIb or IV non-small cell lung cancer HER2 IHC 2+ or 3+ by local laboratory assessment.

Exclusion Criteria:

* Major surgery, radiation therapy, or systemic anti-cancer therapy within 28 days of starting study treatment.
* Some types of brain metastases
* Peripheral neuropathy of Grade 2 within 3 weeks prior to the first study therapy
* History of exposure to cumulative doxorubicin dose ≥ 360 mg/meter squared. If another anthracycline or more than one anthracycline has been used, then the cumulative dose must not exceed the equivalent of 360 mg/meter squared of doxorubicin
* History of clinically significant cardiac dysfunction
* Current known active infection with HIV, hepatitis B virus, or hepatitis C virus
* Current severe, uncontrolled systemic disease
* Severe dyspnea at rest, due to complications of advanced malignancy, or requiring supplementary oxygen therapy.
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or other malignancy with a similar expected curative outcome

Patients who participate in the dose escalation segment of the study cannot participate in the expansion segment of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11-21 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose or recommended Phase 2 dose | Up to 14 weeks, from the date of first dose until unacceptable side effects or a dose-limiting toxicity is met.
  Evaluate adverse events and use of concomitant medication use after XMT-1522 doses

SECONDARY OUTCOMES:
Time of maximum observed concentration of XMT-1522 | Daily for one week after first dose; weekly until 21 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1522
Maximum concentration of XMT-1522 | Daily for one week after first dose; weekly until 21 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1522
Area under the concentration curve of the last measurable concentration of XMT-1522 | Daily for one week after first dose; weekly until 21 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1522
Antineoplastic effects of XMT-1522 | Every 6 weeks up to 12 months
  Monitor tumor size
Anti-drug antibody | Before first dose, 21 and 42 days after first dose, and every 42 days until end of study which is estimated to be 100 days (14 weeks) after first dose
  Analyze blood for antibodies to XMT-1522 and neutralizing antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Eric P. Hailman, MD, PhD, Study Director — Mersana Therapeutics, Inc.
Locations (5):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided